CLINICAL TRIAL: NCT03962686
Title: Molecular Mechanisms Implied in Carotid Atherosclerosis and Atherosclerotic Plaque Progression in Patients Normoglycemics vs. Patients With Diabetes Mellitus
Brief Title: Molecular Mechanisms and Carotid Atherosclerosis
Status: Completed | Type: Observational
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Celestino Sardu, clinical professor, University of Campania Luigi Vanvitelli
Other Study IDs: SecondUNI 22.05.2019
Record Dates: First submitted 2019-05-22; First posted 2019-05-24 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Diabetes Mellitus, Type 2; Atherosclerosis of Artery; Atherosclerotic Plaque
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Plaque, Atherosclerotic | interventions — Hydroxymethylglutaryl-CoA Reductase Inhibitors

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — samples of atherosclerotic plaques obtained during revascularization of carotid arteries.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- normoglycemics: In this cohort will be enrolled 30 normoglycemics patients affected by carotid artery atherosclerotic and evidence of atherosclerotic plaque causing an endolumninal stenosis > 60%. These patients will receive a surgical intervention to remove the atherosclerotic plaque and to revascularize the obstructed coronary artery vessel.
- patients with diabetes mellitus (DM) treated with statin: In this cohort will be enrolled 23 DM patients affected by carotid artery atherosclerotic and evidence of atherosclerotic plaque causing an endolumninal stenosis > 60%. These patients will receive a surgical intervention to remove the atherosclerotic plaque and to revascularize the obstructed coronary artery vessel.
- patients with diabetes mellitus (DM) treated with statin plus PCSK9i: In this cohort will be enrolled 20 DM patients affected by carotid artery atherosclerotic and evidence of atherosclerotic plaque causing an endolumninal stenosis > 60%. These patients will receive a surgical intervention to remove the atherosclerotic plaque and to revascularize the obstructed coronary artery vessel. These patients were treated before the surgical intervention by statin therapy daily (n 20) added to PCSK9i, 140 mg twice a month (n 30).
  Interventions: Drug: statin Oral Tablet plus PCSK9i

INTERVENTIONS:
Drug: statin Oral Tablet plus PCSK9i — Patients in the third study cohort will receive for statin oral therapy plus 140 mg twice a month PCSK9i therapy via subcutaneous injection before to practice surgical intervention for carotid artery obstruction.
  Groups: patients with diabetes mellitus (DM) treated with statin plus PCSK9i

SUMMARY:
The role of methylase system and Proprotein convertase subtilisin/kexin type 9 (PCSK9) in the accelerated atherosclerotic progression of diabetic patients is unclear. Authors will evaluate methylase activity and PCSK9 in carotid plaques of asymptomatic diabetic and non diabetic patients, as well as the effect of statin added to PCSK9 inhibitors (PCSK9i) therapy vs. statin alone in diabetic plaques. Plaques will be obtained from 43 type 2 diabetic and 30 non diabetic patients undergoing carotid endarterectomy. Diabetic patients will receive statin therapy (n 23) or statin plus PCSK9i (140 mg of evolocumab; n 20) or placebo (n 23) for 4 months before scheduled endarterectomy. Plaques will be analyzed for macrophages (CD68), T-cells (CD3), inflammatory cells (HLADR), methylase activity, nuclear factor (NF)-KB, tumor necrosis factor (TNF)-alpha, nitrotyrosine, matrix metalloproteinase (MMP) and collagen content (immunohistochemistry and enzyme- linked immunosorbent assay. Authors' study hypothesis is that methylase and PCSK9 over-activity will be associated with enhanced inflammatory reaction and NF-KB expression in diabetic plaques. Secondly, the inhibition of methylase activity in atherosclerotic lesions of diabetic patients by metformin plus SLGT2i might be associated with morphological and compositional characteristics of a potential stable plaque phenotype, possibly by down regulating NF-KB-mediated inflammatory pathways.

DETAILED DESCRIPTION:
Diabetes Mellitus (DM) leads to increased vulnerability for plaque disruption and mediates increased incidence and severity of clinical events. Inflammation, particularly in diabetes, plays a central role in the cascade of events that result in plaque erosion and fissuring. There is emerging evidence that the methylase system might be involved in both initial stage and progression of atherosclerosis. Moreover, the methylase system might be involved in inflammatory/oxidative stress pathway, involved for activation of nuclear factor kappa B (NF-KB), and other proteins linked to over inflammation/oxidative stress. Although it has been demonstrated that diabetes may up regulate these inflammatory/oxidative pathway, still no evidence exists about the potential role of methylase system in the evolution of atherosclerotic plaques of diabetic patients. Conversely, less data have been reported about the possible modulation of these pathways by drugs as PCSK9i. However, in the present study authors hypothesized that by increasing methylase activity, diabetes may enhance the inflammatory potential of atherosclerotic plaques favoring instability, and its relation with the expression of proprotein convertase subtilisin/kexin type 9 (PCSK9). Therefore, authors designed this study to identify differences in inflammatory infiltration as well as methylase activity and PCSK9 expression between carotid plaques of asymptomatic diabetic and non diabetic (normoglycemics) patients. Because experimental and pathological studies suggest that activation of methylase system might control inflammation/oxidative stress, the present study also evaluated the effect of the statin added to PCSK9i (vs. statin alone) on methylase activity and PCSK9 expression in carotid plaques of diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* evidence of carotid artery atherosclerosis with endoluminal stenosis > 60%;
* aged >18 years.
* aged <75 years

Exclusion Criteria:

* insulin dependent DM;
* absence of carotid artery atherosclerosis with endoluminal stenosis > 60%;
* contraindication to receive a carotid artery revascularization treatment;

  --contraindication to receive metformin treatment;
* controindication to receive PCSK9i treatment;
* neoplastic diseases;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population will be divided in 30 normoglycemics patients vs. 46 DM patients. DM patients will be divided in patients previous treated by oral daily statin therapy (23 patients) vs. DM patients (n 20) previous treated by daily statin therapy plus 140 mg twice a month of PCSK9i. All patients will be affected by severe obstructive carotid artery atherosclerosis.
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
methylase status | 12 months
  to evaluate the activity (over vs. hypo activation) of methylase complex in atherosclerotic carotid plaques of normoglycemics vs. DM patients, and of DM patients treated with statin vs. DM patients previous treated by statin plus PCSK9i

CONTACTS AND LOCATIONS:
Locations (1):
- Raffaele Marfella, Naples, Italy

IPD SHARING:
Plan to Share IPD: Undecided